CLINICAL TRIAL: NCT01682369
Title: A Multi-centre, Phase II, Open Labelled Randomised Control Trial to Describe Immune & Transcriptomic Responses to Trivalent Inactivated Vaccine (TIV) & MF59 Adjuvanted Influenza Vaccine (ATIV) in 14 -26 Month Healthy Children
Brief Title: ADITEC FLU STUDY: Understanding the Genetic Basis for Immune Responses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OVG 2012/04; 2012-002443-26 (EudraCT Number)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 a - TIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine TIV (Agrippal) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine TIV (Agrippal)
  V3-(Day V2+1)- Collect blood sample (up to 6.0 ml)
  V4- Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: TIV (Aggripal)
- Group 1 b - TIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine TIV (Agrippal) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine TIV (Agrippal)
  V3-(Day V2+3)- Collect blood sample (up to 6.0 ml)
  V4- Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: TIV (Aggripal)
- Group 1 c - TIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine TIV (Aggripal) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine TIV (Aggripal)
  V3-(Day V2+7)- Collect blood sample (up to 6.0 ml)
  V4- Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: TIV (Aggripal)
- Group 2 a - ATIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine ATIV (Fluad) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine ATIV (Fluad)
  V3- V3(Day V2+1)- Collect blood sample (up to 6.0 ml)
  V4- V4 Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: ATIV (Fluad)
- Group 2 b - ATIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine ATIV (Fluad) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine ATIV (Fluad)
  V3- V3(Day V2+3)- Collect blood sample (up to 6.0 ml)
  V4- V4 Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: ATIV (Fluad)
- Group 2 c - ATIV (Other): V1- Day 0- Administer a dose of 0.25ml of vaccine ATIV (Fluad) + Collect blood sample (up to 6.0 ml)
  V2- Day 28 (26-35)- Vaccination 2nd dose, Administer a dose of 0.25ml of vaccine ATIV (Fluad)
  V3- V3(Day V2+7)- Collect blood sample (up to 6.0 ml)
  V4- V4 Day V2+28 (26-35)- Collect blood sample (up to 6.0 ml)
  Interventions: Biological: ATIV (Fluad)

INTERVENTIONS:
Biological: TIV (Aggripal)
  Other Names: Begripal
  Arms: Group 1 a - TIV; Group 1 b - TIV; Group 1 c - TIV
Biological: ATIV (Fluad)
  Arms: Group 2 a - ATIV; Group 2 b - ATIV; Group 2 c - ATIV

SUMMARY:
Infants and young children do not respond as well as adults to the flu vaccines currently available in the UK. Fluad, is a different type of influenza vaccine that has been available in the European continent for the last decade, and contains an adjuvant known as MF59.

This vaccine has been used extensively in adults over 65 years of age. It has been administered to over 4000 children in previous studies, which have shown that it produces an enhanced immune response in children compared with traditional vaccines, and that it is safe in this age group. It is, however, not yet licensed for use in children. The reason for this new study is to gain a better understanding of the how this vaccine is stimulating the immune system, by looking to see which parts of the genetic code are 'switched on' in response to immunisation, and to see how this differs from the response to currently used flu vaccines.

To do this the Oxford Vaccine Group will enrol children aged 14 to 26 months to receive either the influenza vaccine with the MF59 adjuvant (ATIV) or one of the influenza vaccines currently available in the UK (Agrippal/ Begripal or TIV). The study will also help to find out whether it is possible to identify patterns of genetic response which can predict responses to immunisation. Being able to do so could potentially enable more rapid development of vaccines against influenza and other diseases in the future. We will also measure how well the immune system responds to the two vaccines and look at any side effects.

The study is funded by Aditec is a collaborative research programme that aims to accelerate the development of novel and powerful immunisation technologies for the next generation of human vaccines.

ELIGIBILITY:
Inclusion Criteria:

* The investigator believes that the parents / LAR (s) of the child can and will comply with requirements of the protocol (e.g. completion of diary cards, understanding of study procedure, consent process, availability at visits)
* Written informed consent obtained from parent / LAR (s) of the subject
* Age from 14 months to 26 months (from start of 14 months up to & excluding 27 months of age)
* Subject is healthy as determined by medical history and clinical examination
* Have received the standard UK immunisation schedule

Exclusion Criteria:

* Child in care
* Use or planned use of any non-registered or investigational product in last 30 days
* Previous influenza vaccination
* Microbiologically proven influenza illness or treatment with antiviral medications
* Confirmed or suspected egg allergy.
* Chronic serious medical conditions which may, in the opinion of the investigator, interfere with evaluation of study objectives e.g. Chronic lung disease, chronic liver/renal disease, chronic renal failure chronic heart disease, congenital genetic syndromes (e.g. Trisomy 21).
* Suspected or confirmed immunosuppressive or immunodeficiency conditions (including splenic dysfunction & HIV)
* Autoimmune conditions e.g. Type 1/2 diabetes mellitus, thyroid disease, juvenile idiopathic arthritis etc.
* Bleeding disorders

Ages: 14 Months to 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Descriptive analyses of gene expression profiles of participants following immunisation with TIV or ATIV in relation to baseline profiles. | 56 days
  To describe gene expression profiles of participants following immunisation with TIV or ATIV in relation to baseline profiles.

SECONDARY OUTCOMES:
To describe the immunogenicity of TIV & ATIV in terms of haemagglutination-Inhibition test (HAI) against each of the three vaccine strains (A/H1N1, A/H3N2, B), four weeks after completion of vaccination. | 56 days
To evaluate the reactogenicity & safety of ATIV in terms of local & systemic reactions following vaccination. | 56 days
To study T&B cell responses following immunisation with each vaccine. | 56 days
To explore the relationship between gene expression and the T cell, B cell and HIA response to immunisation with TIV and ATIV. | 56 days
To explore the relationship between gene expression and the reactogenicity of TIV and ATIV. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — Oxford Vaccine Group; Matthew Snape, PhD, Principal Investigator — Oxford Vaccine Group
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Nakaya HI, Clutterbuck E, Kazmin D, Wang L, Cortese M, Bosinger SE, Patel NB, Zak DE, Aderem A, Dong T, Del Giudice G, Rappuoli R, Cerundolo V, Pollard AJ, Pulendran B, Siegrist CA. Systems biology of immunity to MF59-adjuvanted versus nonadjuvanted trivalent seasonal influenza vaccines in early childhood. Proc Natl Acad Sci U S A. 2016 Feb 16;113(7):1853-8. doi: 10.1073/pnas.1519690113. Epub 2016 Jan 11. PMID 26755593
- See also: OVG website — http://www.ovg.ox.ac.uk